CLINICAL TRIAL: NCT06504914
Title: Developing FIM-BCS: A Lifestyle Modification for African-American Breast Cancer Survivors With Cardiovascular Risk Factors
Brief Title: Preparing FIM-BCS - A Lifestyle Modification for African-American Breast Cancer Survivors
Acronym: FIM-BCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0966
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Obesity; Nutrition, Healthy
MeSH Terms: conditions — Hypertension; Obesity

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arms (Experimental): Participants will attend a 8 week intervention that includes cooking classes, grocery delivery and nutrition education.
  Interventions: Behavioral: Assigned Interventions

INTERVENTIONS:
Behavioral: Assigned Interventions — Behavioral: RN-CHeFRx The RN-CHeFRx trial to enhance dietary intake and blood pressure control in Black women with hypertension and obesity compared to usual care.

SUMMARY:
Hypertension and obesity are both major risk factors for cardiovascular disease (CVD), a leading cause of death for Black women in the United States. The investigators propose examining the feasibility and acceptability of the 12-week RN-CHeFRx (Real Nourishment and Cooking Healthy Food is Rx) intervention

- grocery delivery, cooking classes, and nutrition education - for Black women with hypertension and obesity to improve nutritious eating habits and blood pressure control.

DETAILED DESCRIPTION:
The objective of this study is to conduct the RN-CHeFRx (Real Nourishment and Cooking Healthy Food is Rx) for 12 weeks among Black women who are obese and hypertensive living Chicago. We propose to 1) Pilot the RN-CHEFRx intervention and measures that will be used to assess blood pressure, BMI status, and sodium intake with 20 Black women diagnosed with hypertension and BMI ≥ 30. We will assess the efficacy of the evaluation tools to be used in a future clinical trial at three-time points (baseline, 12 weeks, and 6 months); and 2) Assess the feasibility and acceptability of the RN-CHeFRx intervention using interviews, surveys, and documentary analysis. Findings from this study will inform a larger efficacy trial of RN-CHeFRx to improve dietary behaviors and blood pressure control among Black women with hypertension and obesity

ELIGIBILITY:
Inclusion Criteria:

* self-identified as Black or of African descent
* female
* ≥ 18 years old
* baseline blood pressure ≥130/85 or diagnosed with hypertension and/or BMI ≥ 25

Exclusion Criteria:

* inability to cook in their homes
* cognitive deficits impeding the ability to participate or provide informed consent
* current treatment for cancer
* liver or renal disease
* pregnancy
* lack of English language proficiency

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete the 8 week intervention | [Time Frame: Up to 8 weeks]
  Completion will be measured by class attendance

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No